CLINICAL TRIAL: NCT02978326
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of SAGE-217 in the Treatment of Adult Female Subjects With Severe Postpartum Depression
Brief Title: A Study to Evaluate SAGE-217 in Participants With Severe Postpartum Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-PPD-201
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Postpartum Depression
Keywords: Postpartum Care
MeSH Terms: conditions — Depression, Postpartum | interventions — zuranolone; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: SAGE-217 15/20 mg Oral Solution (Experimental): Participants received SAGE-217, 15 milligrams (mg), oral solution, twice daily (BID) for first 2 days followed by SAGE-217, 15 or 20 mg, oral solution, BID, starting on Day 3 for up to 14 days as tolerated.
  Interventions: Drug: SAGE-217 15/20 mg Oral Solution
- Part B: Placebo (Placebo Comparator): Participants received SAGE-217 matching placebo, capsules, orally, once daily, for up to 14 days.
  Interventions: Drug: Placebo
- Part B: SAGE 217 30 mg Capsules (Experimental): Participants received SAGE-217, 30 mg, capsules, orally, once daily, for up to 14 days.
  Interventions: Drug: SAGE 217 30 mg Capsules

INTERVENTIONS:
Drug: SAGE-217 15/20 mg Oral Solution — SAGE-217, 15 mg oral solution, BID for Days 1 to 2 followed by 20 mg oral solution BID for Days 3 to 14. If not tolerated, 15 mg for the rest of study (Days 3 to 14).
  Arms: Part A: SAGE-217 15/20 mg Oral Solution
Drug: Placebo — SAGE-217 matching placebo, capsules, orally, once daily, for up to 14 days.
  Arms: Part B: Placebo
Drug: SAGE 217 30 mg Capsules — SAGE-217, 30 mg, capsules, orally, once daily, for up to 14 days.
  Arms: Part B: SAGE 217 30 mg Capsules

SUMMARY:
The primary purpose of this study was to determine if treatment with SAGE-217 reduces depressive symptoms in participants with severe postpartum depression (PPD) compared to placebo as assessed by the change from baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D) total score at Day 15 and to evaluate the safety and tolerability of SAGE-217 compared to placebo as assessed by the incidence of adverse events, vital sign measurements, clinical laboratory evaluations, electrocardiogram (ECG) parameters, and the Columbia Suicide Severity Rating Scale (C-SSRS).

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant either must have ceased lactating at screening or, if still lactating or actively breastfeeding at screening, must agree to temporarily cease giving breast milk to her infant(s)
* Participant has had a Major Depressive Episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 Axis I Disorders (SCID-I)
* Participant was <=six months postpartum.

Key Exclusion Criteria:

* Active psychosis
* Attempted suicide associated with current episode of postpartum depression
* Medical history of seizures
* Medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.

Note: suicidal ideation was not an exclusion. Other protocol-defined inclusion/exclusion criteria might apply.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 276 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Sage Investigational Site, Little Rock, Arkansas
  - Sage Investigational Site, Beverly Hills, California
  - Sage Investigational Site, Oceanside, California
  - Sage Investigational Site, Wildomar, California
  - Sage Investigational Site, Washington D.C., District of Columbia
  - Sage Investigational Site, Aventura, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational SIte, Pinellas Park, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Hoffman Estates, Illinois
  - Sage Investigational Site, Owensboro, Kentucky
  - Sage Investigational Site, Lake Charles, Louisiana
  - Sage Investigational Site, New Orleans, Louisiana
  - Sage Investigational Site, Saint Charles, Missouri
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, Manhasset, New York
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Raleigh, North Carolina
  - Sage Investigational Site, Providence, Rhode Island
  - Sage Investigational Site, Fort Worth, Texas
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Richardson, Texas
  - Sage Investigational Site, Orem, Utah

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Result] Deligiannidis K, Lasser R, Gunduz-Bruce H, Silber C, Sankoh AJ, Li Si, et al. A Phase 3, Double-Blind, Placebo- Controlled Trial of SAGE-217 in Postpartum Depression: Assessment of Depressive Symptoms Across Multiple Measures. Abstract presented at: American Society of Clinical Psychopharmacology 2019 Annual Meeting; May 28-31, 2019; Scottsdale, AZ.
- [Result] Lasser R, Deligiannidis K, Gunduz-Bruce H, Silber C, Sankoh AJ, Li Si, et al. A Phase 3, Double-Blind, Placebo- Controlled Trial of SAGE-217 in Postpartum Depression: Topline Assessment of Secondary Efficacy Measures of Anxiety and Depression. Abstract presented at: American Society of Clinical Psychopharmacology 2019 Annual Meeting; May 28-31, 2019; Scottsdale, AZ.
- [Result] Deligiannidis KM, Meltzer-Brody S, Gunduz-Bruce H, Doherty J, Jonas J, Li S, Sankoh AJ, Silber C, Campbell AD, Werneburg B, Kanes SJ, Lasser R. Effect of Zuranolone vs Placebo in Postpartum Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Sep 1;78(9):951-959. doi: 10.1001/jamapsychiatry.2021.1559. PMID 34190962
- [Derived] Deligiannidis KM, Citrome L, Huang MY, Acaster S, Fridman M, Bonthapally V, Lasser R, Kanes SJ. Effect of Zuranolone on Concurrent Anxiety and Insomnia Symptoms in Women With Postpartum Depression. J Clin Psychiatry. 2023 Jan 30;84(1):22m14475. doi: 10.4088/JCP.22m14475. PMID 36724109
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 27 investigative centers in the United States of America from 04 January 2017 to 11 December 2018. Study was conducted in 2 parts. In Part A, only 1 participant was enrolled and thus no analysis was performed for Part A. All analysis sets were defined only for Part B. For Part A, only adverse events incidence were captured.
Pre-assignment Details: A total of 276 participants were enrolled and consented of which 154 eligible participants were randomized and thus presented in participant flow. Rest of the 123 participants were not randomized and not part of any analyses. 152 randomized participants received study drug and 143 completed the study.
Period: Part A (Up to 75 Days)
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Started | 1 | 0 | 0
Completed (Completed = Number of participants who completed Part A of the study.) | 1 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B (Up to 45 Days)
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Started (Started = Number of participants who were randomized to receive study drug in Part B of the study.) | 0 | 76 | 77
Received Study Drug (Two participants were randomized but did not receive study drug (1 in each treatment group).) | 0 | 73 | 78 (Two participants were randomized to placebo but received at least 1 dose of SAGE-217 in error and were included in the SAGE-217 group for 'Received Study Drug' and for 'Safety Analysis'.)
Safety Set (Part B) (Safety Set (Part B) included all participants who were administered study drug in Part B and summarized by actual treatment received.) | 0 | 73 | 78
Efficacy Set (Part B) (Efficacy Set (Part B) included all participants who were administered study drug, had a valid Baseline and at least 1 post-baseline efficacy assessment.) | 0 | 74 | 76
Completed | 0 | 69 | 73
Not Completed | 0 | 7 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Non-compliance | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Part A: All randomized participants; Part B: Efficacy Set included all participants who were administered study drug, had a valid Baseline and at least 1 post-baseline efficacy assessment.
Groups:
- Part A: SAGE-217 15/20 mg Oral Solution: Participants received SAGE-217, 15 mg, oral solution, BID for first 2 days followed by SAGE-217, 15 or 20 mg, oral solution, BID, starting on Day 3 for up to 14 days as tolerated.
- Total: Total of all reporting groups
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules | Total
Number analyzed (Participants) | 1 | 74 | 76 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 74 | 76 | 151
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 74 | 76 | 151
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled during Part A of the study, 0 participants are reported due to the risk of identification of a person.
  Participants
    number analyzed (Participants) | 0 | 74 | 76 | 150
    Hispanic or Latino |  | 18 | 16 | 34
    Not Hispanic or Latino |  | 56 | 60 | 116
    Unknown or Not Reported |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled during Part A of the study, 0 participants are reported due to the risk of identification of a person.
  Participants
    number analyzed (Participants) | 0 | 74 | 76 | 150
    American Indian or Alaska Native |  | 0 | 0 | 0
    Asian |  | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander |  | 1 | 0 | 1
    Black or African American |  | 31 | 31 | 62
    White |  | 40 | 44 | 84
    More than one race |  | 1 | 0 | 1
    Unknown or Not Reported |  | 0 | 0 | 0
17-Item Hamilton Rating Scale for Depression (HAM-D) Total Score [Mean (Full Range); unit: score on a scale] — The 17-item HAM-D is used to rate the severity of depression in participants who are already diagnosed as depressed. Items scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. HAM-D total score=sum of the 17 individual item scores and could range from 0 to 52. Higher scores indicated more severe depression. Population: Only 1 participant was enrolled and treated in the Part A: SAGE-217 15/20 mg Oral Solution arm group and due to low number of participants, no efficacy analyses were conducted for Part A of the study.
  score on a scale
    number analyzed (Participants) | 0 | 74 | 76 | 150
    (all) |  | 28.8 [26 to 40] | 28.4 [26 to 34] | 28.6 [26 to 40]
HAM-D Subscales Scores [Mean (Full Range); unit: score on a scale] — HAM-D is used to rate the severity of depression in participants who are already diagnosed as depressed. HAM-D subscales: Core subscale; Anxiety subscale; Bech-6 subscale; Meier subscale. Each item in the subscale was scored in a range of 0 to 2 or 0 to 4, higher scores=greater degree of depression. Subscale scores were calculated as the sum of the individual item scores comprising each subscale. Scores were transformed to a scale of 0 to 100, with higher scores indicating more severe depression. Population: Only 1 participant was enrolled and treated in the Part A: SAGE-217 15/20 mg Oral Solution arm group and due to low number of participants, no efficacy analyses were conducted for Part A of the study.
  score on a scale
    Core: number analyzed (Participants) | 0 | 74 | 76 | 150
    Core |  | 50.1 [40 to 80] | 51.3 [40 to 70] | 50.7 [40 to 80]
    Anxiety: number analyzed (Participants) | 0 | 74 | 76 | 150
    Anxiety |  | 56.3 [28 to 78] | 53.1 [39 to 78] | 54.7 [28 to 78]
    Bech-6: number analyzed (Participants) | 0 | 74 | 76 | 150
    Bech-6 |  | 64.5 [50 to 86] | 66.3 [50 to 82] | 65.4 [50 to 86]
    Meier: number analyzed (Participants) | 0 | 74 | 76 | 150
    Meier |  | 57.1 [46 to 79] | 59.1 [42 to 83] | 58.1 [42 to 83]
HAM-D Individual Item Scores [Mean (Full Range); unit: score on a scale] — The 17-item HAM-D is used to rate the severity of depression in participants who are already diagnosed as depressed. Individual items on the scale were scored in a range of 0 to 2 or 0 to 4. Symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Symptoms scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Higher scores indicated a greater degree of depression. Population: Only 1 participant was enrolled and treated in the Part A: SAGE-217 15/20 mg Oral Solution arm group and due to low number of participants, no efficacy analyses were conducted for Part A of the study.
  score on a scale
    Depressed Mood: number analyzed (Participants) | 0 | 74 | 76 | 150
    Depressed Mood |  | 3.1 [2 to 4] | 3.1 [3 to 4] | 3.1 [2 to 4]
    Feelings of Guilt: number analyzed (Participants) | 0 | 74 | 76 | 150
    Feelings of Guilt |  | 2.2 [1 to 3] | 2.5 [1 to 3] | 2.35 [1 to 3]
    Suicide: number analyzed (Participants) | 0 | 74 | 76 | 150
    Suicide |  | 0.4 [0 to 3] | 0.4 [0 to 2] | 0.4 [0 to 3]
    Insomnia Early - Early Night: number analyzed (Participants) | 0 | 74 | 76 | 150
    Insomnia Early - Early Night |  | 1.8 [0 to 2] | 1.8 [0 to 2] | 1.8 [0 to 2]
    Insomnia Middle - Middle Night: number analyzed (Participants) | 0 | 74 | 76 | 150
    Insomnia Middle - Middle Night |  | 1.9 [1 to 2] | 1.7 [0 to 2] | 1.8 [0 to 2]
    Insomnia Early Hours - Morning: number analyzed (Participants) | 0 | 74 | 76 | 150
    Insomnia Early Hours - Morning |  | 1.5 [0 to 2] | 1.6 [0 to 2] | 1.55 [0 to 2]
    Work and Activities: number analyzed (Participants) | 0 | 74 | 76 | 150
    Work and Activities |  | 3.1 [1 to 4] | 3.0 [2 to 4] | 3.05 [1 to 4]
    Retardation: number analyzed (Participants) | 0 | 74 | 76 | 150
    Retardation |  | 1.2 [0 to 3] | 1.2 [0 to 3] | 1.2 [0 to 3]
    Agitation: number analyzed (Participants) | 0 | 74 | 76 | 150
    Agitation |  | 1.4 [0 to 3] | 1.4 [0 to 4] | 1.4 [0 to 4]
    Anxiety Psychic: number analyzed (Participants) | 0 | 74 | 76 | 150
    Anxiety Psychic |  | 2.7 [2 to 4] | 2.9 [1 to 4] | 2.8 [1 to 4]
    Anxiety Somatic: number analyzed (Participants) | 0 | 74 | 76 | 150
    Anxiety Somatic |  | 1.9 [0 to 3] | 1.9 [0 to 3] | 1.9 [0 to 3]
    Somatic Symptoms Gastrointestinal: number analyzed (Participants) | 0 | 74 | 76 | 150
    Somatic Symptoms Gastrointestinal |  | 1.5 [0 to 2] | 1.3 [0 to 2] | 1.4 [0 to 2]
    General Somatic Symptoms: number analyzed (Participants) | 0 | 74 | 76 | 150
    General Somatic Symptoms |  | 1.8 [1 to 2] | 1.8 [0 to 2] | 1.8 [0 to 2]
    Genital Symptoms: number analyzed (Participants) | 0 | 74 | 76 | 150
    Genital Symptoms |  | 1.9 [1 to 2] | 1.9 [0 to 2] | 1.9 [0 to 2]
    Hypochondriasis: number analyzed (Participants) | 0 | 74 | 76 | 150
    Hypochondriasis |  | 1.3 [0 to 3] | 1.0 [0 to 3] | 1.15 [0 to 3]
    Loss of Weight According to Patient: number analyzed (Participants) | 0 | 74 | 76 | 150
    Loss of Weight According to Patient |  | 0.9 [0 to 2] | 0.6 [0 to 2] | 0.75 [0 to 2]
    Insight: number analyzed (Participants) | 0 | 74 | 76 | 150
    Insight |  | 0.1 [0 to 1] | 0.1 [0 to 1] | 0.1 [0 to 1]
Montgomery and Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Full Range); unit: score on a scale] — The MADRS is a 10-item questionnaire used to measure the severity of depressive episodes in participants with mood disorders. It includes questions on the following symptoms: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; and suicidal thoughts. Each item was scored in a range of 0 (no symptoms) to 6 (symptoms of maximum severity). MADRS total score was calculated as sum of the 10 individual item scores and could range from 0 to 60. Higher scores indicated more severe depression. Population: Only 1 participant was enrolled and treated in the Part A: SAGE-217 15/20 mg Oral Solution arm group and due to low number of participants, no efficacy analyses were conducted for Part A of the study.
  score on a scale
    number analyzed (Participants) | 0 | 74 | 76 | 150
    (all) |  | 36.3 [27 to 50] | 34.9 [26 to 45] | 35.6 [26 to 50]
Hamilton Anxiety Rating Scale (HAM-A) Total Score [Mean (Full Range); unit: score on a scale] — The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each of the 14 items was defined by a series of symptoms and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The individual items were scored in a range of 0 (not present) to 4 (very severe). The HAM-A total score was calculated as the sum of the 14 individual item scores and could range from 0 to 56 where a score of <17=mild severity; 18-24= mild to moderate severity and 25-30=moderate to severe severity Population: Only 1 participant was enrolled and treated in the Part A: SAGE-217 15/20 mg Oral Solution arm group and due to low number of participants, no efficacy analyses were conducted for Part A of the study.
  score on a scale
    number analyzed (Participants) | 0 | 74 | 76 | 150
    (all) |  | 27.2 [17 to 40] | 26.1 [14 to 40] | 26.65 [14 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Parts A and B: Change From Baseline in the 17-Item Hamilton Rating Scale for Depression (HAM-D) Total Score at Day 15
Description: The 17-item HAM-D is used to rate the severity of depression in participants who are already diagnosed as depressed. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The HAM-D total score was calculated as the sum of the 17 individual item scores and could range from 0 to 52. Higher scores indicated more severe depression. A negative change from Baseline indicates less depression.
Time Frame: Parts A and B: Baseline, Day 15
Population: Only 1 participant was enrolled and treated in the Part A: SAGE-217 15/20 mg Oral Solution arm group and due to low number of participants, no efficacy analyses were conducted for Part A of the study. Part B: Efficacy Set included all participants who were administered study drug, had a valid Baseline and at least 1 post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
score on a scale |  | -13.6 (1.07) | -17.8 (1.04)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Test type: Superiority; p = 0.0028, Mixed Model for Repeated Measures — Mixed Model for Repeated Measures (MMRM) was used for estimation with treatment, baseline HAM-D total score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction as fixed effects; Least Squares (LS) Mean Difference = -4.2, 95% CI 2-sided [-6.9 to -1.5], Standard Error of Mean 1.37

2. Secondary Outcome: Parts A and B: Change From Baseline in the HAM-D Total Score at Days 3, 8, 21 and 45
Description: as for outcome 1
Time Frame: Part B: Baseline, Days 3, 8, 21 and 45
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
score on a scale
  Change From Baseline at Day 3 |  | -9.8 (0.95) | -12.5 (0.93)
  Change From Baseline at Day 8 |  | -12.9 (1.03) | -16.3 (1.00)
  Change From Baseline at Day 21 |  | -14.4 (1.11) | -17.6 (1.09)
  Change From Baseline at Day 45 |  | -15.1 (1.06) | -19.2 (1.02)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change From Baseline in the HAM-D Total Score at Day 3; Test type: Superiority; p = 0.0252, Mixed Model for Repeated Measures — MMRM was used for estimation with treatment, baseline HAM-D total score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction as fixed effects; LS Mean Difference = -2.7, 95% CI 2-sided [-5.1 to -0.3], Standard Error of Mean 1.19
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change From Baseline in the HAM-D Total Score at Day 8; Test type: Superiority; p = 0.0106, Mixed Model for Repeated Measures — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -3.4, 95% CI 2-sided [-6.0 to -0.8], Standard Error of Mean 1.31
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change From Baseline in the HAM-D Total Score at Day 21; Test type: Superiority; p = 0.0321, Mixed Model for Repeated Measures — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -3.1, 95% CI 2-sided [-6.0 to -0.3], Standard Error of Mean 1.44
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change From Baseline in the HAM-D Total Score at Day 45; Test type: Superiority; p = 0.0027, Mixed Model for Repeated Measures — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -4.1, 95% CI 2-sided [-6.7 to -1.4], Standard Error of Mean 1.34

3. Secondary Outcome: Parts A and B: Percentage of Participants With HAM-D Response
Description: HAM-D Response was defined as having a 50 percent (%) or greater reduction from Baseline in HAM-D total score. The HAM-D total score was calculated as the sum of the 17 individual item scores and could range from 0 to 52. The items on HAM-D included: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early night, middle night, early hours [morning]), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Higher scores indicated more depression.
Time Frame: Part B: Days 3, 8, 15, 21 and 45
Population: Only 1 participant was enrolled and treated in the Part A: SAGE-217 15/20 mg Oral Solution arm group and due to low number of participants, no efficacy analyses were conducted for Part A of the study. Part B: Efficacy Set included all participants who were administered study drug, had a valid Baseline and at least 1 post-baseline efficacy assessment. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
percentage of participants
  Day 3: number analyzed (Participants) | 0 | 74 | 74
  Day 3 |  | 27.0 | 40.5
  Day 8: number analyzed (Participants) | 0 | 74 | 75
  Day 8 |  | 44.6 | 65.3
  Day 15: number analyzed (Participants) | 0 | 73 | 74
  Day 15 |  | 47.9 | 71.6
  Day 21: number analyzed (Participants) | 0 | 73 | 74
  Day 21 |  | 56.2 | 71.6
  Day 45: number analyzed (Participants) | 0 | 69 | 73
  Day 45 |  | 56.5 | 75.3
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Response at Day 3; Test type: Superiority; p = 0.1004, GEE for binary response model — Generalized estimating equations (GEE) for binary response model was used for estimation with factors for treatment, baseline HAM-D total score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.89 to 3.60]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Response at Day 8; Test type: Superiority; p = 0.0127, GEE for binary response model — Generalized estimating equations for binary response model was used for estimation with factors for treatment, baseline HAM-D total score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.20 to 4.45]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Response at Day 15; Test type: Superiority; p = 0.0049, GEE for binary response model — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.34 to 5.16]
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Response at Day 21; Test type: Superiority; p = 0.0763, GEE for binary response model — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.94 to 3.64]
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Response at Day 45; Test type: Superiority; p = 0.0216, GEE for binary response model — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.13 to 4.60]

4. Secondary Outcome: Parts A and B: Percentage of Participants With HAM-D Remission
Description: HAM-D Remission was defined as a HAM-D total score of less than or equal to (<=)7. The HAM-D total score was calculated as the sum of the 17 individual item scores and could range from 0 to 52. The items on HAM-D included: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early night, middle night, early hours [morning]), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Higher scores indicated more depression.
Time Frame: Part B: Days 3, 8, 15, 21 and 45
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
percentage of participants
  Day 3: number analyzed (Participants) | 0 | 74 | 74
  Day 3 |  | 5.4 | 18.9
  Day 8: number analyzed (Participants) | 0 | 74 | 75
  Day 8 |  | 18.9 | 32.0
  Day 15: number analyzed (Participants) | 0 | 73 | 74
  Day 15 |  | 23.3 | 44.6
  Day 21: number analyzed (Participants) | 0 | 73 | 74
  Day 21 |  | 28.8 | 41.9
  Day 45: number analyzed (Participants) | 0 | 69 | 73
  Day 45 |  | 30.4 | 53.4
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Remission at Day 3; Test type: Superiority; p = 0.0200, GEE for binary response model — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 3.89, 95% CI 2-sided [1.24 to 12.23]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Remission at Day 8; Test type: Superiority; p = 0.0990, GEE for binary response model — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.89 to 4.13]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Remission at Day 15; Test type: Superiority; p = 0.0110, GEE for binary response model — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.24 to 5.17]
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Remission at Day 21; Test type: Superiority; p = 0.1982, GEE for binary response model — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.79 to 3.19]
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With HAM-D Remission at Day 45; Test type: Superiority; p = 0.0091, GEE for binary response model — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 2.52, 95% CI 2-sided [1.26 to 5.03]

5. Secondary Outcome: Parts A and B: Change From Baseline in HAM-D Subscales Scores
Description: HAM-D is used to rate the severity of depression in participants who are already diagnosed as depressed. HAM-D subscales: Core subscale (symptoms-depressed mood, feelings of guilt, suicide, work and activities, and retardation ); Anxiety subscale (symptoms-anxiety [psychic and somatic], somatic symptoms [gastrointestinal and general], hypochondriasis, loss of weight); Bech-6 subscale (symptoms-depressed mood, feelings of guilt, work and activities, retardation, anxiety psychic, and somatic symptoms general); Meier subscale (symptoms-depressed mood, feelings of guilt, work and activities, retardation, agitation, and anxiety psychic). Each item was scored in a range of 0 to 2 or 0 to 4, higher scores=greater degree of depression. Subscale scores were calculated as the sum of the individual item scores comprising each subscale. Scores were transformed to a scale of 0 to 100, with higher scores indicated more severe depression. A negative change from Baseline indicates less depression.
Time Frame: Part B: Baseline, Days 3, 8, 15, 21 and 45
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
score on a scale
  Core: Change From Baseline at Day 3 |  | -16.7 (1.91) | -18.8 (1.88)
  Core: Change From Baseline at Day 8 |  | -23.4 (2.03) | -28.7 (1.99)
  Core: Change From Baseline at Day 15 |  | -26.8 (2.10) | -31.9 (2.06)
  Core: Change From Baseline at Day 21 |  | -27.3 (2.24) | -33.7 (2.20)
  Core: Change From Baseline at Day 45 |  | -29.5 (2.11) | -37.2 (2.05)
  Anxiety: Change From Baseline at Day 3 |  | -16.4 (1.98) | -23.5 (1.93)
  Anxiety: Change From Baseline at Day 8 |  | -23.2 (2.15) | -29.8 (2.09)
  Anxiety: Change From Baseline at Day 15 |  | -23.4 (2.19) | -33.2 (2.13)
  Anxiety: Change From Baseline at Day 21 |  | -27.3 (2.17) | -33.3 (2.11)
  Anxiety: Change From Baseline at Day 45 |  | -26.5 (2.19) | -34.5 (2.11)
  Bech-6: Change From Baseline at Day 3 |  | -19.5 (2.45) | -23.7 (2.41)
  Bech-6: Change From Baseline at Day 8 |  | -28.3 (2.58) | -34.9 (2.53)
  Bech-6: Change From Baseline at Day 15 |  | -30.9 (2.61) | -39.2 (2.56)
  Bech-6: Change From Baseline at Day 21 |  | -32.7 (2.72) | -40.7 (2.68)
  Bech-6: Change From Baseline at Day 45 |  | -34.6 (2.61) | -44.0 (2.54)
  Meier: Change From Baseline at Day 3 |  | -17.0 (2.17) | -21.7 (2.13)
  Meier: Change From Baseline at Day 8 |  | -25.0 (2.30) | -32.2 (2.24)
  Meier: Change From Baseline at Day 15 |  | -28.1 (2.35) | -35.5 (2.30)
  Meier: Change From Baseline at Day 21 |  | -29.9 (2.42) | -37.0 (2.37)
  Meier: Change From Baseline at Day 45 |  | -31.5 (2.32) | -41.0 (2.25)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Core: Change from Baseline in HAM-D Subscale Score at Day 3; Test type: Superiority; p = 0.3832, Mixed Model for Repeated Measures — MMRM was used for estimation with treatment, baseline HAM-D subscale score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction as fixed effects; LS Mean Difference = -2.1, 95% CI 2-sided [-6.9 to 2.7], Standard Error of Mean 2.41
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Core: Change from Baseline in HAM-D Subscale Score at Day 8; Test type: Superiority; p = 0.0415, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -5.4, 95% CI 2-sided [-10.5 to -0.2], Standard Error of Mean 2.60
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Core: Change from Baseline in HAM-D Subscale Score at Day 15; Test type: Superiority; p = 0.0606, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -5.1, 95% CI 2-sided [-10.5 to 0.2], Standard Error of Mean 2.71
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Core: Change from Baseline in HAM-D Subscale Score at Day 21; Test type: Superiority; p = 0.0318, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -6.3, 95% CI 2-sided [-12.1 to -0.6], Standard Error of Mean 2.91
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Core: Change from Baseline in HAM-D Subscale Score at Day 45; Test type: Superiority; p = 0.0047, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -7.7, 95% CI 2-sided [-13.0 to -2.4], Standard Error of Mean 2.69
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety: Change from Baseline in HAM-D Subscale Score at Day 3; Test type: Superiority; p = 0.0053, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -7.1, 95% CI 2-sided [-12.0 to -2.1], Standard Error of Mean 2.50
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety: Change from Baseline in HAM-D Subscale Score at Day 8; Test type: Superiority; p = 0.0181, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -6.6, 95% CI 2-sided [-12.1 to -1.1], Standard Error of Mean 2.76
Statistical Analysis 8: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety: Change from Baseline in HAM-D Subscale Score at Day 15; Test type: Superiority; p = 0.0007, Mixed Model for Repeated Measures; LS Mean Difference = -9.8, 95% CI 2-sided [-15.3 to -4.2], Standard Error of Mean 2.82
Statistical Analysis 9: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety: Change from Baseline in HAM-D Subscale Score at Day 21; Test type: Other; p = 0.0332, Mixed Model for Repeated Measures; LS Mean Difference = -6.0, 95% CI 2-sided [-11.5 to -0.5], Standard Error of Mean 2.79
Statistical Analysis 10: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety: Change from Baseline in HAM-D Subscale Score at Day 45; Test type: Other; p = 0.0048, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -8.0, 95% CI 2-sided [-13.5 to -2.5], Standard Error of Mean 2.80
Statistical Analysis 11: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Bech-6: Change from Baseline in HAM-D Subscale Score at Day 3; Test type: Superiority; p = 0.1840, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -4.2, 95% CI 2-sided [-10.3 to 2.0], Standard Error of Mean 3.12
Statistical Analysis 12: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Bech-6: Change from Baseline in HAM-D Subscale Score at Day 8; Test type: Superiority; p = 0.0462, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -6.7, 95% CI 2-sided [-13.2 to -0.1], Standard Error of Mean 3.31
Statistical Analysis 13: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Bech-6: Change from Baseline in HAM-D Subscale Score at Day 15; Test type: Superiority; p = 0.0150, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -8.3, 95% CI 2-sided [-14.9 to -1.6], Standard Error of Mean 3.36
Statistical Analysis 14: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Bech-6: Change from Baseline in HAM-D Subscale Score at Day 21; Test type: Superiority; p = 0.0245, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -8.0, 95% CI 2-sided [-15.0 to -1.0], Standard Error of Mean 3.53
Statistical Analysis 15: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Bech-6: Change from Baseline in HAM-D Subscale Score at Day 45; Test type: Superiority; p = 0.0054, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -9.4, 95% CI 2-sided [-16.0 to -2.8], Standard Error of Mean 3.34
Statistical Analysis 16: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Meier: Change from Baseline in HAM-D Subscale Score at Day 3; Test type: Superiority; p = 0.0972, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -4.6, 95% CI 2-sided [-10.1 to 0.9], Standard Error of Mean 2.77
Statistical Analysis 17: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Meier: Change from Baseline in HAM-D Subscale Score at Day 8; Test type: Superiority; p = 0.0155, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -7.2, 95% CI 2-sided [-13.1 to -1.4], Standard Error of Mean 2.95
Statistical Analysis 18: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Meier: Change from Baseline in HAM-D Subscale Score at Day 15; Test type: Superiority; p = 0.0149, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -7.5, 95% CI 2-sided [-13.4 to -1.5], Standard Error of Mean 3.03
Statistical Analysis 19: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Meier: Change from Baseline in HAM-D Subscale Score at Day 21; Test type: Superiority; p = 0.0250, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -7.1, 95% CI 2-sided [-13.3 to -0.9], Standard Error of Mean 3.14
Statistical Analysis 20: Comparison: Part B: Placebo; Meier: Change from Baseline in HAM-D Subscale Score at Day 45; Test type: Superiority; p = 0.0017, Mixed Model for Repeated Measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -9.5, 95% CI 2-sided [-15.3 to -3.6], Standard Error of Mean 2.96

6. Secondary Outcome: Parts A and B: Change From Baseline in HAM-D Individual Item Scores
Description: The 17-item HAM-D is used to rate the severity of depression in participants who are already diagnosed as depressed. Individual items on the scale were scored in a range of 0 to 2 or 0 to 4. Symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms were scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Higher scores indicated a greater degree of depression. A negative change from Baseline indicates less depression.
Time Frame: Part B: Baseline, Days 3, 8, 15, 21 and 45
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
score on a scale
  Depressed Mood: Change From Baseline at Day 3 |  | -0.8 (0.13) | -1.1 (0.13)
  Depressed Mood: Change From Baseline at Day 8 |  | -1.3 (0.14) | -1.7 (0.13)
  Depressed Mood: Change From Baseline at Day 15 |  | -1.5 (0.15) | -1.8 (0.13)
  Depressed Mood: Change From Baseline at Day 21 |  | -1.5 (0.14) | -2.1 (0.13)
  Depressed Mood: Change From Baseline at Day 45 |  | -1.7 (0.15) | -2.1 (0.12)
  Feelings of Guilt: Change From Baseline at Day 3 |  | -0.9 (0.12) | -1.0 (0.13)
  Feelings of Guilt: Change From Baseline at Day 8 |  | -1.1 (0.13) | -1.4 (0.12)
  Feelings of Guilt: Change From Baseline at Day 15 |  | -1.3 (0.13) | -1.5 (0.11)
  Feelings of Guilt: Change From Baseline at Day 21 |  | -1.2 (0.13) | -1.6 (0.12)
  Feelings of Guilt: Change From Baseline at Day 45 |  | -1.5 (0.12) | -1.8 (0.11)
  Suicide: Change From Baseline at Day 3 |  | -0.2 (0.05) | -0.3 (0.04)
  Suicide: Change From Baseline at Day 8 |  | -0.2 (0.04) | -0.4 (0.03)
  Suicide: Change From Baseline at Day 15 |  | -0.3 (0.04) | -0.3 (0.04)
  Suicide: Change From Baseline at Day 21 |  | -0.2 (0.05) | -0.3 (0.05)
  Suicide: Change From Baseline at Day 45 |  | -0.2 (0.05) | -0.4 (0.03)
  Insomnia Early - Early Night: Change From Baseline at Day 3 |  | -0.9 (0.11) | -1.2 (0.10)
  Insomnia Early - Early Night: Change From Baseline at Day 8 |  | -0.9 (0.11) | -1.3 (0.10)
  Insomnia Early - Early Night: Change From Baseline at Day 15 |  | -0.9 (0.11) | -1.3 (0.10)
  Insomnia Early - Early Night: Change From Baseline at Day 21 |  | -0.9 (0.11) | -1.1 (0.10)
  Insomnia Early - Early Night: Change From Baseline at Day 45 |  | -1.0 (0.12) | -1.1 (0.11)
  Insomnia Middle - Middle Night: Change From Baseline at Day 3 |  | -1.0 (0.11) | -1.3 (0.10)
  Insomnia Middle - Middle Night: Change From Baseline at Day 8 |  | -1.0 (0.11) | -1.3 (0.09)
  Insomnia Middle - Middle Night: Change From Baseline at Day 15 |  | -0.9 (0.11) | -1.3 (0.09)
  Insomnia Middle - Middle Night: Change From Baseline at Day 21 |  | -0.8 (0.11) | -1.2 (0.09)
  Insomnia Middle - Middle Night: Change From Baseline at Day 45 |  | -0.9 (0.11) | -1.3 (0.10)
  Insomnia Early Hours - Morning: Change From Baseline at Day 3 |  | -0.8 (0.11) | -1.1 (0.10)
  Insomnia Early Hours - Morning: Change From Baseline at Day 8 |  | -0.9 (0.10) | -1.2 (0.09)
  Insomnia Early Hours - Morning: Change From Baseline at Day 15 |  | -1.0 (0.11) | -1.2 (0.09)
  Insomnia Early Hours - Morning: Change From Baseline at Day 21 |  | -0.9 (0.11) | -1.0 (0.10)
  Insomnia Early Hours - Morning: Change From Baseline at Day 45 |  | -0.9 (0.10) | -1.3 (0.08)
  Work and Activities: Change From Baseline at Day 3 |  | -0.8 (0.12) | -0.9 (0.13)
  Work and Activities: Change From Baseline at Day 8 |  | -1.3 (0.14) | -1.4 (0.14)
  Work and Activities: Change From Baseline at Day 15 |  | -1.4 (0.14) | -1.8 (0.13)
  Work and Activities: Change From Baseline at Day 21 |  | -1.7 (0.16) | -1.9 (0.14)
  Work and Activities: Change From Baseline at Day 45 |  | -1.7 (0.16) | -2.1 (0.14)
  Retardation: Change From Baseline at Day 3 |  | -0.5 (0.07) | -0.4 (0.10)
  Retardation: Change From Baseline at Day 8 |  | -0.7 (0.08) | -0.8 (0.07)
  Retardation: Change From Baseline at Day 15 |  | -0.8 (0.07) | -0.8 (0.07)
  Retardation: Change From Baseline at Day 21 |  | -0.8 (0.08) | -0.8 (0.07)
  Retardation: Change From Baseline at Day 45 |  | -0.9 (0.07) | -1.0 (0.07)
  Agitation: Change From Baseline at Day 3 |  | -0.4 (0.09) | -0.7 (0.09)
  Agitation: Change From Baseline at Day 8 |  | -0.6 (0.09) | -0.9 (0.08)
  Agitation: Change From Baseline at Day 15 |  | -0.6 (0.09) | -0.9 (0.09)
  Agitation: Change From Baseline at Day 21 |  | -0.8 (0.09) | -0.9 (0.08)
  Agitation: Change From Baseline at Day 45 |  | -0.8 (0.09) | -1.1 (0.07)
  Anxiety Psychic: Change From Baseline at Day 3 |  | -0.7 (0.12) | -1.1 (0.13)
  Anxiety Psychic: Change From Baseline at Day 8 |  | -1.1 (0.14) | -1.5 (0.13)
  Anxiety Psychic: Change From Baseline at Day 15 |  | -1.2 (0.13) | -1.6 (0.13)
  Anxiety Psychic: Change From Baseline at Day 21 |  | -1.3 (0.14) | -1.6 (0.12)
  Anxiety Psychic: Change From Baseline at Day 45 |  | -1.3 (0.14) | -1.7 (0.12)
  Anxiety Somatic: Change From Baseline at Day 3 |  | -0.6 (0.10) | -0.7 (0.10)
  Anxiety Somatic: Change From Baseline at Day 8 |  | -0.7 (0.10) | -0.9 (0.10)
  Anxiety Somatic: Change From Baseline at Day 15 |  | -0.8 (0.11) | -0.9 (0.10)
  Anxiety Somatic: Change From Baseline at Day 21 |  | -0.9 (0.11) | -1.0 (0.11)
  Anxiety Somatic: Change From Baseline at Day 45 |  | -0.8 (0.11) | -1.0 (0.10)
  Somatic Symptoms Gastrointestinal: Change From Baseline at Day 3 |  | -0.3 (0.09) | -0.6 (0.10)
  Somatic Symptoms Gastrointestinal: Change From Baseline at Day 8 |  | -0.6 (0.10) | -0.8 (0.09)
  Somatic Symptoms Gastrointestinal: Change From Baseline at Day 15 |  | -0.7 (0.11) | -1.0 (0.08)
  Somatic Symptoms Gastrointestinal: Change From Baseline at Day 21 |  | -0.8 (0.11) | -0.9 (0.09)
  Somatic Symptoms Gastrointestinal: Change From Baseline at Day 45 |  | -0.8 (0.10) | -1.0 (0.09)
  General Somatic Symptoms: Change From Baseline at Day 3 |  | -0.6 (0.08) | -0.7 (0.09)
  General Somatic Symptoms: Change From Baseline at Day 8 |  | -0.8 (0.09) | -0.9 (0.09)
  General Somatic Symptoms: Change From Baseline at Day 15 |  | -0.6 (0.08) | -1.1 (0.09)
  General Somatic Symptoms: Change From Baseline at Day 21 |  | -0.7 (0.10) | -1.0 (0.08)
  General Somatic Symptoms: Change From Baseline at Day 45 |  | -0.8 (0.09) | -1.0 (0.09)
  Genital Symptoms: Change From Baseline at Day 3 |  | -0.3 (0.08) | -0.4 (0.09)
  Genital Symptoms: Change From Baseline at Day 8 |  | -0.6 (0.10) | -0.6 (0.09)
  Genital Symptoms: Change From Baseline at Day 15 |  | -0.7 (0.10) | -0.9 (0.10)
  Genital Symptoms: Change From Baseline at Day 21 |  | -0.7 (0.10) | -0.8 (0.10)
  Genital Symptoms: Change From Baseline at Day 45 |  | -0.8 (0.10) | -1.0 (0.10)
  Hypochondriasis: Change From Baseline at Day 3 |  | -0.5 (0.09) | -0.7 (0.08)
  Hypochondriasis: Change From Baseline at Day 8 |  | -0.6 (0.08) | -0.8 (0.07)
  Hypochondriasis: Change From Baseline at Day 15 |  | -0.5 (0.10) | -1.0 (0.06)
  Hypochondriasis: Change From Baseline at Day 21 |  | -0.6 (0.08) | -0.9 (0.06)
  Hypochondriasis: Change From Baseline at Day 45 |  | -0.7 (0.09) | -0.9 (0.07)
  Loss of Weight According to Patient: Change From Baseline at Day 3 |  | -0.3 (0.08) | -0.5 (0.07)
  Loss of Weight According to Patient: Change From Baseline at Day 8 |  | -0.4 (0.07) | -0.5 (0.07)
  Loss of Weight According to Patient: Change From Baseline at Day 15 |  | -0.5 (0.07) | -0.5 (0.06)
  Loss of Weight According to Patient: Change From Baseline at Day 21 |  | -0.6 (0.06) | -0.6 (0.05)
  Loss of Weight According to Patient: Change From Baseline at Day 45 |  | -0.5 (0.08) | -0.6 (0.05)
  Insight: Change From Baseline at Day 3 |  | 0.0 (0.02) | -0.1 (0.02)
  Insight: Change From Baseline at Day 8 |  | 0.0 (0.02) | -0.1 (0.02)
  Insight: Change From Baseline at Day 15 |  | 0.0 (0.02) | -0.1 (0.02)
  Insight: Change From Baseline at Day 21 |  | 0.0 (0.02) | -0.1 (0.02)
  Insight: Change From Baseline at Day 45 |  | 0.0 (0.04) | -0.1 (0.02)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Depressed Mood: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.1569, Mixed Model for Repeated Measures — MMRM was used for estimation with treatment, baseline HAM-D individual item score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction as fixed effects; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Depressed Mood: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0376, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to 0.0], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Depressed Mood: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.1035, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Depressed Mood: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.0037, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.18
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Depressed Mood: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0061, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.1], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Feelings of Guilt: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.7878, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Feelings of Guilt: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0498, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Feelings of Guilt: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.1719, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Feelings of Guilt: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.0161, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.16
Statistical Analysis 10: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Feelings of Guilt: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0191, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.15
Statistical Analysis 11: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Suicide: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.2537, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.06
Statistical Analysis 12: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Suicide: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0018, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to -0.1], Standard Error of Mean 0.04
Statistical Analysis 13: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Suicide: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.2878, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.05
Statistical Analysis 14: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Suicide: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.2594, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 15: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Suicide: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0086, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.06
Statistical Analysis 16: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early - Early Night: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.0424, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.14
Statistical Analysis 17: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early - Early Night: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0207, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.14
Statistical Analysis 18: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early - Early Night: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0010, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.14
Statistical Analysis 19: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early - Early Night: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.0871, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.14
Statistical Analysis 20: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early - Early Night: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.5680, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.15
Statistical Analysis 21: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Middle - Middle Night: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.0143, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.14
Statistical Analysis 22: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Middle - Middle Night: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0063, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.13
Statistical Analysis 23: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Middle - Middle Night: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0042, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.13
Statistical Analysis 24: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Middle - Middle Night: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.0137, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.13
Statistical Analysis 25: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Middle - Middle Night: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0099, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.14
Statistical Analysis 26: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early Hours - Morning: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.0507, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.14
Statistical Analysis 27: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early Hours - Morning: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0205, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.13
Statistical Analysis 28: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early Hours - Morning: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.1409, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.13
Statistical Analysis 29: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early Hours - Morning: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority — MMRM was used for estimation with treatment, baseline HAM-D individual item score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction as fixed effects; p = 0.2021, Mixed Model for Repeated Measures; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.14
Statistical Analysis 30: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insomnia Early Hours - Morning: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0117, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.12
Statistical Analysis 31: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Work and Activities: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.5511, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.15
Statistical Analysis 32: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Work and Activities: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.4949, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.18
Statistical Analysis 33: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Work and Activities: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0203, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.17
Statistical Analysis 34: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Work and Activities: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.2076, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.19
Statistical Analysis 35: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Work and Activities: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0362, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.8 to 0.0], Standard Error of Mean 0.19
Statistical Analysis 36: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Retardation: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.3589, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.12
Statistical Analysis 37: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Retardation: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.6991, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10
Statistical Analysis 38: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Retardation: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.9655, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10
Statistical Analysis 39: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Retardation: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.8699, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10
Statistical Analysis 40: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Retardation: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.3715, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 41: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Agitation: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.0670, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.12
Statistical Analysis 42: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Agitation: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0104, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.11
Statistical Analysis 43: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Agitation: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0122, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.12
Statistical Analysis 44: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Agitation: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.3157, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.12
Statistical Analysis 45: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Agitation: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0077, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.11
Statistical Analysis 46: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Psychic: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.0078, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.8 to -0.1], Standard Error of Mean 0.16
Statistical Analysis 47: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Psychic: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0372, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to 0.0], Standard Error of Mean 0.18
Statistical Analysis 48: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Psychic: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0244, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.17
Statistical Analysis 49: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Psychic: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.0993, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.17
Statistical Analysis 50: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Psychic: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0185, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.17
Statistical Analysis 51: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Somatic: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.2471, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.12
Statistical Analysis 52: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Somatic: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.1076, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.14
Statistical Analysis 53: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Somatic: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.2782, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.14
Statistical Analysis 54: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Somatic: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.4646, Mixed Model for Repeated Measures; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.15
Statistical Analysis 55: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Anxiety Somatic: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.1600, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.14
Statistical Analysis 56: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Somatic Symptoms Gastrointestinal: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.0474, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.12
Statistical Analysis 57: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Somatic Symptoms Gastrointestinal: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0446, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.12
Statistical Analysis 58: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Somatic Symptoms Gastrointestinal: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0093, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.12
Statistical Analysis 59: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Somatic Symptoms Gastrointestinal: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.2998, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.12
Statistical Analysis 60: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Somatic Symptoms Gastrointestinal: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0545, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.12
Statistical Analysis 61: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; General Somatic Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.2177, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.12
Statistical Analysis 62: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; General Somatic Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.2300, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.12
Statistical Analysis 63: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; General Somatic Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0001, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.12
Statistical Analysis 64: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; General Somatic Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.0151, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.12
Statistical Analysis 65: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; General Somatic Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0502, Mixed Model for Repeated Measures; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.13
Statistical Analysis 66: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Genital Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.3659, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.11
Statistical Analysis 67: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Genital Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.6003, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.12
Statistical Analysis 68: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Genital Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0785, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.13
Statistical Analysis 69: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Genital Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.3668, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.13
Statistical Analysis 70: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Genital Symptoms: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.1827, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.13
Statistical Analysis 71: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Hypochondriasis: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.1327, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.12
Statistical Analysis 72: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Hypochondriasis: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.0993, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.11
Statistical Analysis 73: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Hypochondriasis: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0002, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.11
Statistical Analysis 74: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Hypochondriasis: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.0056, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.10
Statistical Analysis 75: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Hypochondriasis: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0122, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.11
Statistical Analysis 76: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Loss of Weight According to Patient: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.1305, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.10
Statistical Analysis 77: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Loss of Weight According to Patient: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.6638, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 78: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Loss of Weight According to Patient: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.4341, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08
Statistical Analysis 79: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Loss of Weight According to Patient: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.9085, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.07
Statistical Analysis 80: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Loss of Weight According to Patient: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.1820, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.09
Statistical Analysis 81: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insight: Change From Baseline in HAM-D Individual Item Score at Day 3; Test type: Superiority; p = 0.1593, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.03
Statistical Analysis 82: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insight: Change From Baseline in HAM-D Individual Item Score at Day 8; Test type: Superiority; p = 0.6555, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.03
Statistical Analysis 83: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insight: Change From Baseline in HAM-D Individual Item Score at Day 15; Test type: Superiority; p = 0.0170, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.03
Statistical Analysis 84: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insight: Change From Baseline in HAM-D Individual Item Score at Day 21; Test type: Superiority; p = 0.0188, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.03
Statistical Analysis 85: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Insight: Change From Baseline in HAM-D Individual Item Score at Day 45; Test type: Superiority; p = 0.0726, Mixed Model for Repeated Measures — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.05

7. Secondary Outcome: Parts A and B: Change From Baseline in Montgomery and Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item questionnaire used to measure the severity of depressive episodes in participants with mood disorders. It includes questions on the following symptoms: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; and suicidal thoughts. Each item was scored in a range of 0 (no symptoms) to 6 (symptoms of maximum severity). The MADRS total score was calculated as the sum of the 10 individual item scores and could range from 0 to 60. Higher scores indicated more severe depression. A negative change from Baseline indicates less depression.
Time Frame: Part B: Baseline, Days 3, 8, 15, 21 and 45
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
score on a scale
  Change From Baseline at Day 3 |  | -11.7 (1.36) | -14.8 (1.33)
  Change From Baseline at Day 8 |  | -16.3 (1.45) | -20.3 (1.42)
  Change From Baseline at Day 15 |  | -17.6 (1.48) | -22.1 (1.45)
  Change From Baseline at Day 21 |  | -17.8 (1.49) | -22.1 (1.46)
  Change From Baseline at Day 45 |  | -19.0 (1.44) | -24.8 (1.39)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change From Baseline in MADRS Total Score at Day 3; Test type: Superiority; p = 0.0791, Mixed Model for Repeated Measures — MMRM was used for estimation with treatment with treatment, baseline MADRS total score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction as fixed effects; LS Mean Difference = -3.0, 95% CI 2-sided [-6.5 to 0.4], Standard Error of Mean 1.72
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change From Baseline in MADRS Total Score at Day 8; Test type: Superiority; p = 0.0322, Mixed Model for Repeated Measures — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -4.0, 1.86% CI 2-sided [-7.7 to -0.3], Standard Error of Mean 1.86
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change From Baseline in MADRS Total Score at Day 15; Test type: Superiority; p = 0.0180, Mixed Model for Repeated Measures — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -4.6, 95% CI 2-sided [-8.3 to -0.8], Standard Error of Mean 1.91
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change from Baseline in MADRS Total Score at 21; Test type: Superiority; p = 0.0271, Mixed Model for Repeated Measures — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -4.3, 95% CI 2-sided [-8.1 to -0.5], Standard Error of Mean 1.92
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change from Baseline in MADRS Total Score at 45; Test type: Superiority; p = 0.0018, Mixed Model for Repeated Measures — [p-value comment as in outcome 7, analysis 1]; LS Mean Difference = -5.8, 95% CI 2-sided [-9.4 to -2.2], Standard Error of Mean 1.82

8. Secondary Outcome: Parts A and B: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response
Description: The Clinical Global Impression - Improvement (CGI-I) item of the CGI scale uses a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. CGI response was defined as a CGI-I score of 1 (very much improved) or 2 (much improved). The percentage of participants with overall improvement in post-treatment condition, rated by investigator as very much improved (CGI-I score of 1) or much improved (CGI-I score of 2) is reported.
Time Frame: Part B: Days 3, 8, 15, 21 and 45
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
percentage of participants
  Day 3: number analyzed (Participants) | 0 | 74 | 74
  Day 3 |  | 28.4 | 37.8
  Day 8: number analyzed (Participants) | 0 | 74 | 75
  Day 8 |  | 50.0 | 65.3
  Day 15: number analyzed (Participants) | 0 | 73 | 74
  Day 15 |  | 52.1 | 71.6
  Day 21: number analyzed (Participants) | 0 | 73 | 74
  Day 21 |  | 54.8 | 70.3
  Day 45: number analyzed (Participants) | 0 | 68 | 73
  Day 45 |  | 55.9 | 71.2
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With CGI-I Response at Day 3; Test type: Superiority; p = 0.3372, GEE for binary response model — Generalized estimating equations for binary response model was used for estimation with factors for treatment, baseline CGI-S score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.70 to 2.81]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With CGI-I Response at Day 8; Test type: Superiority; p = 0.0935, GEE for binary response model — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.91 to 3.47]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With CGI-I Response at Day 15; Test type: Superiority; p = 0.0276, GEE for binary response model — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.09 to 4.28]
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With CGI-I Response at Day 21; Test type: Superiority; p = 0.0920, GEE for binary response model — Generalized estimating equations for binary response model was used for estimation with factors for treatment: Baseline CGI-S score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.91 to 3.54]
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With CGI-I Response at Day 45; Test type: Superiority; p = 0.1109, GEE for binary response model — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.88 to 3.51]

9. Secondary Outcome: Parts A and B: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score
Description: The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each of the 14 items was defined by a series of symptoms and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The individual items were scored in a range of 0 (not present) to 4 (very severe). The HAM-A total score was calculated as the sum of the 14 individual item scores and could range from 0 to 56 where a score of <17=mild severity; 18-24= mild to moderate severity and 25-30=moderate to severe severity. A negative change from Baseline indicates less anxiety.
Time Frame: Part B: Baseline, Days 3, 8, 15, 21 and 45
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
score on a scale
  Change From Baseline at Day 3 |  | -8.9 (1.02) | -12.0 (0.99)
  Change From Baseline at Day 8 |  | -11.7 (1.04) | -16.1 (1.01)
  Change From Baseline at Day 15 |  | -12.7 (1.09) | -16.6 (1.07)
  Change From Baseline at Day 21 |  | -13.1 (1.07) | -16.6 (1.05)
  Change From Baseline at Day 45 |  | -13.6 (1.02) | -18.6 (0.99)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change from Baseline in HAM-A Total Score at Day 3; Test type: Superiority; p = 0.0169, Mixed Model for Repeated Measures — MMRM was used for estimation with treatment, baseline HAM-A total score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction as fixed effects; LS Mean Difference = -3.1, 95% CI 2-sided [-5.7 to -0.6], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change from Baseline in HAM-A Total Score at Day 8; Test type: Superiority; p = 0.0010, Mixed Model for Repeated Measures — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -4.4, 95% CI 2-sided [-7.0 to -1.8], Standard Error of Mean 1.32
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change from Baseline in HAM-A Total Score at Day 15; Test type: Superiority; p = 0.0063, Mixed Model for Repeated Measures — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -3.9, 95% CI 2-sided [-6.7 to -1.1], Standard Error of Mean 1.41
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change from Baseline in HAM-A Total Score at Day 21; Test type: Superiority; p = 0.0119, Mixed Model for Repeated Measures — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -3.5, 95% CI 2-sided [-6.2 to -0.8], Standard Error of Mean 1.37
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Change from Baseline in HAM-A Total Score at Day 45; Test type: Superiority; p = 0.0002, Mixed Model for Repeated Measures — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -5.0, 95% CI 2-sided [-7.5 to -2.4], Standard Error of Mean 1.28

10. Secondary Outcome: Parts A and B: Percentage of Participants With MADRS Response
Description: MADRS response was defined as having a 50% or greater reduction from Baseline in MADRS total score. The MADRS is a 10-item questionnaire used to measure the severity of depressive episodes in participants with mood disorders. It includes questions on the following symptoms: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; and suicidal thoughts. Each item was scored in a range of 0 (no symptoms) to 6 (symptoms of maximum severity). The MADRS total score was calculated as the sum of the 10 individual item scores and could range from 0 to 60. Higher scores indicated more depression.
Time Frame: Part B: Days 3, 8, 15, 21 and 45
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
percentage of participants
  Day 3: number analyzed (Participants) | 0 | 74 | 74
  Day 3 |  | 27.0 | 40.5
  Day 8: number analyzed (Participants) | 0 | 74 | 75
  Day 8 |  | 50.0 | 64.0
  Day 15: number analyzed (Participants) | 0 | 73 | 74
  Day 15 |  | 47.9 | 73.0
  Day 21: number analyzed (Participants) | 0 | 73 | 74
  Day 21 |  | 52.1 | 70.3
  Day 45: number analyzed (Participants) | 0 | 69 | 73
  Day 45 |  | 56.5 | 74.0
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Response at Day 3; Test type: Superiority; p = 0.1145, GEE for binary response model — Generalized estimating equations for binary response model was used for estimation with factors for treatment, baseline MADRS total score, baseline antidepressant use, assessment time point, and time point-by-treatment interaction; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.87 to 3.53]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Response at Day 8; Test type: Superiority; p = 0.1069, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.89 to 3.30]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Response at Day 15; Test type: Superiority; p = 0.0045, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.36 to 5.27]
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Response at Day 21; Test type: Superiority; p = 0.0421, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.03 to 3.93]
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Response at Day 45; Test type: Superiority; p = 0.0541, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.99 to 4.03]

11. Secondary Outcome: Parts A and B: Percentage of Participants With MADRS Remission
Description: MADRS Remission was defined as a MADRS total score of <=10. The MADRS is a 10-item questionnaire used to measure the severity of depressive episodes in participants with mood disorders. It includes questions on the following symptoms: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; and suicidal thoughts. Each item was scored in a range of 0 (no symptoms) to 6 (symptoms of maximum severity). The MADRS total score was calculated as the sum of the 10 individual item scores and could range from 0 to 60. Higher scores indicated more depression.
Time Frame: Part B: Days 3, 8, 15, 21 and 45
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 0 | 74 | 76
percentage of participants
  Day 3: number analyzed (Participants) | 0 | 74 | 74
  Day 3 |  | 9.5 | 24.3
  Day 8: number analyzed (Participants) | 0 | 74 | 75
  Day 8 |  | 28.4 | 37.3
  Day 15: number analyzed (Participants) | 0 | 73 | 74
  Day 15 |  | 30.1 | 54.1
  Day 21: number analyzed (Participants) | 0 | 73 | 74
  Day 21 |  | 31.5 | 52.7
  Day 45: number analyzed (Participants) | 0 | 69 | 73
  Day 45 |  | 37.7 | 58.9
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Remission at Day 3; Test type: Superiority; p = 0.0326, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.09 to 7.38]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Remission at Day 8; Test type: Superiority; p = 0.3749, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.68 to 2.79]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Remission at Day 15; Test type: Superiority; p = 0.0087, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.49, 95% CI 2-sided [1.26 to 4.92]
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Remission at Day 21; Test type: Superiority; p = 0.0257, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.10 to 4.31]
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: SAGE 217 30 mg Capsules; Percentage of Participants With MADRS Remission at Day 45; Test type: Superiority; p = 0.0339, GEE for binary response model — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.06 to 4.09]

12. Secondary Outcome: Parts A and B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an AE with an onset that occurs after receiving study drug.
Time Frame: Part A: Up to Day 75; Part B: Up to Day 45
Population: Part A: All randomized participants; Part B: Safety Set included all participants who were administered study drug in Part B of the study and analyzed as per actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 1 | 73 | 78
Participants | 1 | 38 | 47

13. Secondary Outcome: Part B: Number of Participants With Potentially Clinically Significant Vital Sign Measurements
Description: Vital signs included assessments of supine and standing systolic blood pressure (SBP), supine and standing diastolic blood pressure (DBP), and heart rate.
Time Frame: Part B: From first dose of study drug up to 45 days
Population: Safety Set (Part B) included all participants who were administered study drug in Part B of the study and analyzed by treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 73 | 78
Participants
  Supine SBP: <90 millimeter of mercury (mmHg) | 0 | 3
  Supine SBP: Decrease From Baseline of >=30 | 2 | 1
  Supine SBP: Increase From Baseline of >=30 | 1 | 0
  Standing SBP: <90 mmHg | 5 | 4
  Standing SBP: Decrease From Baseline of >=30 | 4 | 1
  Standing SBP: Increase From Baseline of >=30 | 1 | 2
  Supine DBP: <50 mmHg | 1 | 1
  Supine DBP: Decrease From Baseline of >=20 | 5 | 3
  Supine DBP: Increase From Baseline of >=20 | 1 | 5
  Standing DBP: <50 mmHg | 1 | 1
  Standing DBP: >110 mmHg | 0 | 1
  Standing DBP: Decrease From Baseline of >=20 | 3 | 7
  Standing DBP: Increase From Baseline of >=20 | 3 | 4

14. Secondary Outcome: Part B: Number of Participants With Potentially Clinically Significant Laboratory Evaluations
Description: Laboratory tests included tests of Hematology, Chemistry, and Urinalysis.
Time Frame: Part B: From first dose of study drug up to 45 days
Population: Safety Set (Part B) included all participants who were administered study drug in Part B and analyzed by treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 73 | 78
Participants
  Hematology: Eosinophils >1.5 10^9/Liter(L) | 0 | 1
  Hematology: Hematocrit <0.359 | 11 | 8
  Hematology: Hematocrit >0.446 | 10 | 12
  Hematology: Hemoglobin <110 g/L | 12 | 6
  Hematology: Leukocytes <2.5 10^9/L | 2 | 2
  Hematology: Neutrophils <1.5 10^9/L | 15 | 11
  Serum Chemistry: Alanine Aminotransferase >3xUpper Limit of Normal Value (ULN) | 1 | 0
  Serum Chemistry: Calcium <2.0 millimoles (mmol)/L | 0 | 1
  Serum Chemistry: Chloride <90 mmol/L | 1 | 2
  Serum Chemistry: Glucose <2.8 mmol/L | 0 | 1
  Serum Chemistry: Glucose >13.9 mmol/L | 0 | 1
  Serum Chemistry: Phosphate >5 milligrams/deciliter (mg/dL) | 2 | 1
  Serum Chemistry: Potassium <3.5 mmol/L | 0 | 1
  Serum Chemistry: Potassium >5.2 mmol/L | 6 | 5
  Serum Chemistry: Sodium >145 mmol/L | 3 | 5

15. Secondary Outcome: Part B: Change From Baseline in Electrocardiogram (ECG) Parameter Heart Rate
Description: ECG parameters included assessment of the standard 12-lead ECG intervals: QT, QTcF, PR, RR, QRS, and heart rate. Heart rate was measured in terms of beats per minute. Change from Baseline in heart rate at specified time points were reported.
Time Frame: Part B: Baseline, Days 8, 15, and 21
Population: Safety Set (Part B) included all participants who were administered study drug in Part B and analyzed by treatment actually received. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 73 | 78
beats per minute
  Baseline | 68.2 (9.55) | 69.9 (10.85)
  Change From Baseline at Day 8: number analyzed (Participants) | 72 | 76
  Change From Baseline at Day 8 | 0.8 (9.91) | 1.5 (12.62)
  Change From Baseline at Day 15: number analyzed (Participants) | 71 | 75
  Change From Baseline at Day 15 | -0.1 (8.16) | 0.9 (12.69)
  Change From Baseline at Day 21: number analyzed (Participants) | 71 | 76
  Change From Baseline at Day 21 | 2.5 (8.93) | -0.6 (11.33)

16. Secondary Outcome: Part B: Change From Baseline in ECG Parameters-PR Interval, RR Interval, QRS Duration, QT Interval, QTcF Interval
Description: ECG parameters included assessment of the standard 12-lead ECG intervals: QT, QTcF, PR, RR, QRS, and heart rate. Change from Baseline in PR Interval, RR Interval, QRS Duration, QT Interval, QTcF Interval is reported.
Time Frame: Part B: Baseline, Days 8, 15, and 21
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 73 | 78
milliseconds
  PR Interval: Baseline: number analyzed (Participants) | 72 | 78
  PR Interval: Baseline | 151.4 (20.38) | 151.7 (17.12)
  PR Interval: Change From Baseline at Day 8: number analyzed (Participants) | 71 | 76
  PR Interval: Change From Baseline at Day 8 | 3.4 (26.97) | 0.6 (11.95)
  PR Interval: Change From Baseline at Day 15: number analyzed (Participants) | 70 | 75
  PR Interval: Change From Baseline at Day 15 | 1.1 (11.81) | 0.8 (11.02)
  PR Interval: Change From Baseline at Day 21: number analyzed (Participants) | 70 | 76
  PR Interval: Change From Baseline at Day 21 | 2.5 (14.66) | 2.5 (11.82)
  RR Interval: Baseline | 892.2 (131.63) | 871.6 (124.16)
  RR Interval: Change From Baseline at Day 8: number analyzed (Participants) | 72 | 76
  RR Interval: Change From Baseline at Day 8 | -9.9 (137.12) | -16.9 (149.42)
  RR Interval: Change From Baseline at Day 15: number analyzed (Participants) | 71 | 75
  RR Interval: Change From Baseline at Day 15 | -1.9 (107.37) | -8.4 (147.36)
  RR Interval: Change From Baseline at Day 21: number analyzed (Participants) | 71 | 76
  RR Interval: Change From Baseline at Day 21 | -32.0 (113.89) | 13.9 (141.69)
  QRS Duration: Baseline | 87.3 (9.50) | 90.2 (9.81)
  QRS Duration: Change From Baseline at Day 8: number analyzed (Participants) | 72 | 76
  QRS Duration: Change From Baseline at Day 8 | 0.0 (8.19) | -0.3 (6.98)
  QRS Duration: Change From Baseline at Day 15: number analyzed (Participants) | 71 | 75
  QRS Duration: Change From Baseline at Day 15 | -0.7 (7.14) | -0.3 (6.69)
  QRS Duration: Change From Baseline at Day 21: number analyzed (Participants) | 71 | 76
  QRS Duration: Change From Baseline at Day 21 | 0.1 (7.58) | 0.0 (6.84)
  QT Interval: Baseline | 395.1 (28.85) | 393.0 (28.66)
  QT Interval: Change From Baseline at Day 8: number analyzed (Participants) | 72 | 76
  QT Interval: Change From Baseline at Day 8 | -5.5 (24.23) | -4.3 (29.89)
  QT Interval: Change From Baseline at Day 15: number analyzed (Participants) | 71 | 75
  QT Interval: Change From Baseline at Day 15 | -1.4 (22.96) | -2.7 (28.53)
  QT Interval: Change From Baseline at Day 21: number analyzed (Participants) | 71 | 76
  QT Interval: Change From Baseline at Day 21 | -5.9 (23.70) | 0.1 (30.60)
  QTcF Interval: Baseline | 411.3 (20.92) | 412.2 (18.83)
  QTcF Interval: Change From Baseline at Day 8: number analyzed (Participants) | 72 | 76
  QTcF Interval: Change From Baseline at Day 8 | -4.1 (15.80) | -1.7 (15.57)
  QTcF Interval: Change From Baseline at Day 15: number analyzed (Participants) | 71 | 75
  QTcF Interval: Change From Baseline at Day 15 | -1.2 (14.75) | -1.5 (14.94)
  QTcF Interval: Change From Baseline at Day 21: number analyzed (Participants) | 71 | 76
  QTcF Interval: Change From Baseline at Day 21 | -1.1 (19.39) | -1.8 (20.77)

17. Secondary Outcome: Part B: Number of Participants With a Response of "Yes" to Any Suicidal Ideation or Suicidal Behaviors Item Using the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS was used to assess the suicidality of participants during the study. The assessment included "yes" or "no" responses for 5 questions, each related to suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Numeric ratings were provided for severity of ideation (if present), from 1 to 5, with 5 being the most severe. Number of participants with a response of 'yes' to any suicidal ideation or suicidal behavior item as measured by C-SSRS is reported.
Time Frame: Part B: Up to Day 45
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
Number analyzed (Participants) | 73 | 78
Participants
  Suicidal Ideation | 13 | 6
  Suicidal Behavior | 0 | 0

ADVERSE EVENTS:
Time Frame: Part A: Up to Day 75; Part B: Up to Day 45
Description: Part A: All randomized participants; Part B: Safety Set included all participants who were administered study drug in Part B of the study and analyzed as per actual treatment received.
Arm/Group | Part A: SAGE-217 15/20 mg Oral Solution | Part B: Placebo | Part B: SAGE 217 30 mg Capsules
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/73 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/73 | 1/78
Other Adverse Events (participants affected / at risk) | 1/1 | 26/73 | 31/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAGE-217 15/20 mg Oral Solution (N=1) | Part B: Placebo (N=73) | Part B: SAGE 217 30 mg Capsules (N=78)
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAGE-217 15/20 mg Oral Solution (N=1) | Part B: Placebo (N=73) | Part B: SAGE 217 30 mg Capsules (N=78)
Somnolence (Nervous system disorders) | 0 | 8 | 12
Headache (Nervous system disorders) | 0 | 9 | 7
Dizziness (Nervous system disorders) | 0 | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 5
Sedation (Nervous system disorders) | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 6 | 3
Vomiting (Gastrointestinal disorders) | 0 | 4 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT02978326/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02978326/SAP_001.pdf